CLINICAL TRIAL: NCT05859399
Title: The Effect of Laughter Yoga on Premenstrual Symptoms and Quality of Life in Midwifery Students With Premenstrual Syndrome
Brief Title: The Effect of Laughter Yoga on Premenstrual Symptoms and Quality of Life in Midwifery Students
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Ahu AKSOY, Research Assistant, PhD, Mersin University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 001
Record Dates: First submitted 2023-05-05; First posted 2023-05-16 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Premenstrual Syndrome; Quality of Life
Keywords: Premenstrual Syndrome; Quality of life; Laughter yoga; Laughter therapy; Student
MeSH Terms: conditions — Premenstrual Syndrome | interventions — Laughter Therapy

STUDY DESIGN:
Intervention Model Description: Prospective, parallel, two arm, randomized controlled clinical trial
Who Masked: Outcomes Assessor
Masking Description: Statistical analysis of the data will be done by an expert independent of the research.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (laughter yoga) group (Experimental): The intervention group will receive 12 online laughter yoga sessions, only one session per week for 12 weeks. In this study, the number of laughter yoga sessions was determined in line with the studies in the literature. Each laughter yoga session is planned to last approximately 40-45 minutes. Each session of laughter yoga consists of clapping and warm-up exercises, deep breathing exercises, childlike play and laughter.
  Interventions: Other: Laughter yoga
- Control group (No Intervention): The control group will receive no intervention for 12 weeks.

INTERVENTIONS:
Other: Laughter yoga — Although the history of laughter yoga dates back to ancient times, its use in medicine has become widespread in the 21st century, while it is used to reduce pain, anxiety, stress, depression and fatigue, it is also a method that can be used to accelerate immunity, quality of life, happiness, sleep quality and recovery.
  Other Names: Laughter therapy
  Arms: Experimental (laughter yoga) group

SUMMARY:
The research was planned as a prospective, randomized controlled experimental study to determine the effect of laughter yoga applied to midwifery students on premenstrual symptoms (PMS) and quality of life.

Research Hypotheses H0: Online laughter yoga has no effect on premenstrual symptoms. H1: Online laughter yoga has an effect on premenstrual symptoms. H0: Online laughter yoga has no effect on quality of life. H1: Online laughter yoga has an impact on quality of life.

DETAILED DESCRIPTION:
59 midwifery students will participate in the research. In this study, the number of laughter yoga sessions was determined in line with the studies in the literature. Each laughter yoga session is planned to last approximately 40-45 minutes. Each session of laughter yoga consists of clapping and warm-up exercises, deep breathing exercises, childlike play and laughter.

ELIGIBILITY:
Inclusion Criteria:

* To agree to participate in the research,
* To be over 18 years old,
* Not having taken vocational courses
* Not having a chronic disease,
* Having a regular menstrual period,
* Having at least 110 points on the PMS scale
* Not receiving medical treatment for PMS.

Exclusion Criteria:

* Refusing to participate in the research,
* To have taken vocational courses,
* Having a chronic illness
* Getting a score lower than 110 on the PMS scale,
* Having any condition where laughter yoga should be avoided (having had abdominal surgery in the last three months, taking regular medications, epilepsy, uncontrollable hypertension, glaucoma, hernia, etc.)
* Receiving medical treatment for PMS.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 58 (Estimated)
Dates: Start 2023-05-15 (Estimated); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Premenstrual Syndrome Scale (PMSS) | change from baseline, at the end of 12th week of intervention.
  The Premenstrual Syndrome Scale is a five-point Likert type scale consisting of 44 questions that measures the severity of premenstrual symptoms, based on DSM-III and DSM-IV-R, in order to measure the severity of premenstrual symptoms

SECONDARY OUTCOMES:
World Health Organization Quality of Life Instrument, Short Form (WHOQOL-BREF) | change from baseline, at the end of 12th week of intervention.
  Life of quality will be evaluated by using the WHOQOL-BREF-TR. This scale consists of 27 questions. There are a total of five areas in the scale: physical, mental, social, environmental and national environmental areas. Each area is evaluated within itself. The domain score is calculated with the score it gets from the questions that determine it. Field scores are evaluated between 4-20. Increasing score indicates goodness.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The effect of online laughter therapy on depression, anxiety, stress, and loneliness among nursing students during the Covid-19 pandemic — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC9477613/pdf/main.pdf